CLINICAL TRIAL: NCT06879483
Title: Early and Intermediate Term Outcomes of Thoraco-laparoscopic Partial Esophagogastrectomy for Management of Esophageal Cancer
Brief Title: Thoraco-laparoscopic Partial Esophagogastrectomy for Management of Esophageal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous Salaheldin, assisstant lecturer of general surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-2-5MD
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thoraco-laparoscopic partial esophagogastrectomy (Experimental): Patients diagnosed with resectable esophageal cancer will undergo thoraco-laparoscopic partial esophagogastrectomy
  Interventions: Procedure: Thoraco-laparoscopic partial esophagogastrectomy

INTERVENTIONS:
Procedure: Thoraco-laparoscopic partial esophagogastrectomy — 1. Laparoscopic Phase:
     * The stomach is mobilized, and a part of it is resected to include the lower esophageal segment.
     * Left gastric nodes, the splenic and common hepatic nodes are dissected.
     * A gastric tube is created using endoscopic staplers for esophageal reconstruction and fixed to the proximal gastrectomy specimen using sutures
  2. Thoracoscopic Phase:
     * The patient is positioned in prone position
     * Three small incisions are made in the thorax
     * Further esophageal mobilization through a right thoracoscopy is performed in left lateral decubitus. Periesophageal nodes are retrieved en bloc. Left and right paratracheal and subcarinal lymph nodes are resected separately. The esophagus is transected at the tumor's proximal margin.
  3. Reconstruction:
     * An anastomosis (esophagogastric connection) is performed to restore continuity, typically using a circular stapler or hand-sewn technique.

SUMMARY:
Thoraco-laparoscopic partial esophagogastrectomy has emerged as a promising minimally invasive alternative, combining thoracoscopy and laparoscopy to reduce the trauma associated with open surgery.Early and intermediate-term outcomes provide critical information on both the oncological efficacy and functional benefits of the procedure. By examining recurrence rates within the first 12-24 months, this study will provide valuable insights into the oncological robustness of this approach compared to more invasive approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with resectable esophageal cancer (stages I-III).
* Suitable for thoraco-laparoscopic partial esophagogastrectomy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Presence of distant metastasis at diagnosis.
* History of previous esophageal or gastric surgery.
* Contraindications to laparoscopy or thoracoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Immediate Postoperative complications | first month post operative
  30-day morbidity and mortality (using Clavien-Dindo classification)
Dysphagia | Collected at base line preoperative,one month, and 12 months post-surgery.
  yes or no
resection margin status | 2 weeks postoperative
  resection margin status (R0/R1/R2)
lymph node yield. | first month post operative
  number of lymph nodes in specimen
regurgitation | Collected at one month, and 12 months post-surgery.
  yes or no

SECONDARY OUTCOMES:
recurrence rate | first year post operative
body mass index | Collected at base line preoperative,one month, and 12 months post-surgery.
serum albumin | Collected at base line preoperative,one month, and 12 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided